CLINICAL TRIAL: NCT04970225
Title: Functional and Phenotypic Characteristics of Blood Neutrophils in Cystic Fibrosis
Brief Title: Cystic Fibrosis Blood Neutrophils
Acronym: MUCO-PNN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: APHP180430; 2018-A03017-48 (Other: ID-RCB Number)
Record Dates: First submitted 2019-01-17; First posted 2021-07-21 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Cystic Fibrosis
Keywords: Blood neutrophils; Pseudomonas aeruginosa; Cystic fibrosis; CFTR modulators; respiratory exacerbation; airway chronic infection
MeSH Terms: conditions — Cystic Fibrosis; Pseudomonas Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Stable state (Experimental): 45 adult cystic fibrosis patients followed in the respiratory medicine department of Cochin hospital, paris, France:
  * With severe cftr mutations
  * With or without PA chronic infection
  * Treated or not with Ivacaftor-Lumacaftor
  Interventions: Other: 1 blood sample
- Starting Ivacaftor-Tezacaftor-Elexacaftor (Experimental): 40 adult cystic fibrosis patients followed in the respiratory medicine department of Cochin hospital, paris, France:
  * With at least one severe cftr mutation
  * With or without PA chronic infection
  * Initiating Ivacaftor-Tezacaftor-Elexacaftor
  Interventions: Other: 2 blood samples
- Exacerbation (Experimental): 15 adult cystic fibrosis patients followed in the respiratory medicine department of Cochin hospital, paris, France and hospitalized for respiratory exacerbation
  Interventions: Other: 2 blood samples

INTERVENTIONS:
Other: 1 blood sample — 4 tubes of 7 ml per sample (a single sample)
  Arms: Stable state
Other: 2 blood samples — 4 tubes of 7 ml per sample / 2 samples : before / after antibiotic treatment
  Arms: Exacerbation; Starting Ivacaftor-Tezacaftor-Elexacaftor

SUMMARY:
The purpose of this prospective study is to analyze function and phenotype of blood neutrophils in cystic fibrosis patients and the impact of Pseudomonas aeruginosa chronic infection, treatment with CFTR modulators and acute exacerbation on blood neutrophils phenotype and function.

ELIGIBILITY:
Inclusion Criteria:

* Patient over the age of 18 who is not under legal protection
* Patients with CF according to the diagnostic criteria of the Cystic Fibrosis Foundation including:

  * 15 patients with severe mutation but not chronically infected with PA and not treated with lumacaftor / ivacaftor
  * 15 patients homozygous phe508del, chronically infected with PA and not treated with lumacaftor / ivacaftor
  * 15 patients homozygous phe508del, chronically infected with PA and treated with lumacaftor / ivacaftor
  * 15 hospitalized patients for respiratory exacerbation
  * 40 patients initiating Ivacaftor-Tezacaftor-Elexacaftor treatment.
* No change in baseline treatment for 15 days (including antibiotic treatment).
* Patient affiliated to a social security system
* Free, informed and written consent, dated and signed by the patient and the investigator, at the latest on the day of inclusion and before any action required by the study.

Exclusion Criteria:

* Informed consent impossible to obtain
* Involvement in an interventional research protocol in the previous 3 months if exclusion directive was given in this protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2021-07-08 (Actual); Primary Completion 2023-04-06 (Actual); Study Completion 2025-01-08 (Actual)

PRIMARY OUTCOMES:
Quantification of blood low density neutrophils in cystic fibrosis (CF) | Through study completion, an average of 1 year
  Quantitative flow cytometric evaluation of neutrophil membrane markers that differ according to whether they are :
  * mature neutrophils : CD16high, CD15high, CD33high, CD10high
  * or Low density neutrophils (LDG) : CD16low, CD15neg, CD33 neg, CD10 neg. Comparison of neutrophil membrane markers profile in CF patients versus control blood-donors.
Transcriptomic analysis of blood neutrophils in cystic fibrosis (CF) | Through study completion, an average of 1 year
  Transcriptomic analysis of blood neutrophil proinflammatory or immunomodulatory potential.
  Comparison of transcriptomic blood neutrophil profile in CF patients versus control blood-donors.
Effector function analysis of blood neutrophils in CF. | Through study completion, an average of 1 year
  Comparison of effector function analysis of blood neutrophils of CF patients versus control blood-donors.
Phagocytosis potential of blood neutrophils in CF. | Through study completion, an average of 1 year
  Comparison of phagocytosis potential of blood neutrophils of CF patients versus control blood-donors.
Survival/apoptosis balance analysis in CF | Through study completion, an average of 1 year
  Survival / apoptosis balance analysis : (PCNA localization) in CF patients blood neutrophils versus control blood-donors.

SECONDARY OUTCOMES:
Quantification of blood low density neutrophils in CF vs other chronic inflammatory disorders. | Through study completion, an average of 1 year
  Quantitative flow cytometric evaluation of neutrophil membrane markers that differ according to whether they are:
  * mature neutrophils : CD16high, CD15high, CD33high, CD10high
  * Low density neutrophils (LDG) : CD16low, CD15neg, CD33 neg, CD10 neg. Comparison of neutrophil membrane markers profile in CF patients versus patients with other chronic inflammatory disease (eg. Rheumatoid arthritis, inflammatory bowel disease).
Quantification of blood low density neutrophils in CF according to different clinical situations. | Through study completion, an average of 1 year
  Quantitative flow cytometric evaluation of neutrophil membrane markers.
  * At stable state:
    * presence or absence of airway chronic infection with PA
    * whether or not patients are treated Ivacaftor-Lumacaftor
  * At beginning of exacerbation or after antibiotic treatment.
  * Before or after Ivacaftor-Tezacaftor-Elexacaftor treatment
Transcriptomic analysis of blood neutrophils in CF according to different clinical situations. | Through study completion, an average of 1 year
  Transcriptomic analysis of blood neutrophil proinflammatory or immunomodulatory potential.
  * At stable state:
    * presence or absence of airway chronic infection with PA
    * whether or not patients are treated Ivacaftor-Lumacaftor
  * At beginning of exacerbation or after antibiotic treatment.
  * Before or after Ivacaftor-Tezacaftor-Elexacaftor treatment
Effector function analysis of blood neutrophils in CF according to different clinical situations. | Through study completion, an average of 1 year
  Effector function analysis of blood neutrophils:
  * At stable state:
    * presence or absence of airway chronic infection with PA
    * whether or not patients are treated Ivacaftor-Lumacaftor
  * At beginning of exacerbation or after antibiotic treatment.
  * Before or after Ivacaftor-Tezacaftor-Elexacaftor treatment
Phagocytosis potential of blood neutrophils in CF according to different clinical situations. | Through study completion, an average of 1 year
  Phagocytosis potential analysis of blood neutrophils in CF:
  * At stable state:
    * presence or absence of airway chronic infection with PA
    * whether or not patients are treated Ivacaftor-Lumacaftor
  * At beginning of exacerbation or after antibiotic treatment.
  * Before or after Ivacaftor-Tezacaftor-Elexacaftor treatment
Survival/apoptosis balance analysis in CF according to different clinical situations. | Through study completion, an average of 1 year
  Survival / apoptosis balance analysis (PCNA localization):
  * At stable state:
    * presence or absence of airway chronic infection with PA
    * whether or not patients are treated Ivacaftor-Lumacaftor
  * At beginning of exacerbation or after antibiotic treatment.
  * Before or after Ivacaftor-Tezacaftor-Elexacaftor treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-Régis BURGEL, MD PHD, Principal Investigator — APHP
Locations (1):
- Cochin hospital, AP-HP, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wright R, Keller G, Gould SJ, Subramani S, Rine J. Cell-type control of membrane biogenesis induced by HMG-CoA reductase. New Biol. 1990 Oct;2(10):915-21. PMID 2078559
- [Background] Bonvillain RW, Painter RG, Adams DE, Viswanathan A, Lanson NA Jr, Wang G. RNA interference against CFTR affects HL60-derived neutrophil microbicidal function. Free Radic Biol Med. 2010 Dec 15;49(12):1872-80. doi: 10.1016/j.freeradbiomed.2010.09.012. Epub 2010 Sep 24. PMID 20870018
- [Background] Bouayad D, Pederzoli-Ribeil M, Mocek J, Candalh C, Arlet JB, Hermine O, Reuter N, Davezac N, Witko-Sarsat V. Nuclear-to-cytoplasmic relocalization of the proliferating cell nuclear antigen (PCNA) during differentiation involves a chromosome region maintenance 1 (CRM1)-dependent export and is a prerequisite for PCNA antiapoptotic activity in mature neutrophils. J Biol Chem. 2012 Sep 28;287(40):33812-25. doi: 10.1074/jbc.M112.367839. Epub 2012 Jul 30. PMID 22846997
- [Background] Bruijnzeel PL, Uddin M, Koenderman L. Targeting neutrophilic inflammation in severe neutrophilic asthma: can we target the disease-relevant neutrophil phenotype? J Leukoc Biol. 2015 Oct;98(4):549-56. doi: 10.1189/jlb.3VMR1214-600RR. Epub 2015 May 14. PMID 25977288
- [Background] Bulloch MN, Hanna C, Giovane R. Lumacaftor/ivacaftor, a novel agent for the treatment of cystic fibrosis patients who are homozygous for the F580del CFTR mutation. Expert Rev Clin Pharmacol. 2017 Oct;10(10):1055-1072. doi: 10.1080/17512433.2017.1378094. Epub 2017 Sep 22. PMID 28891346
- [Background] Chiara AD, Pederzoli-Ribeil M, Burgel PR, Danel C, Witko-Sarsat V. Targeting cytosolic proliferating cell nuclear antigen in neutrophil-dominated inflammation. Front Immunol. 2012 Oct 9;3:311. doi: 10.3389/fimmu.2012.00311. eCollection 2012. PMID 23181059
- [Background] Cantin A. Cystic fibrosis lung inflammation: early, sustained, and severe. Am J Respir Crit Care Med. 1995 Apr;151(4):939-41. doi: 10.1164/ajrccm.151.4.7697269. No abstract available.
- [Background] Vaz WL, Nisksch A, Jahnig F. Electrostatic interactions at charged lipid membranes. Measurement of surface pH with fluorescent lipoid pH indicators. Eur J Biochem. 1978 Feb 1;83(1):299-305. doi: 10.1111/j.1432-1033.1978.tb12094.x. PMID 23947
- [Background] Downey DG, Bell SC, Elborn JS. Neutrophils in cystic fibrosis. Thorax. 2009 Jan;64(1):81-8. doi: 10.1136/thx.2007.082388. PMID 19103874
- [Background] Fadok VA, Bratton DL, Henson PM. Phagocyte receptors for apoptotic cells: recognition, uptake, and consequences. J Clin Invest. 2001 Oct;108(7):957-62. doi: 10.1172/JCI14122. No abstract available. PMID 11581295
- [Background] Futosi K, Mocsai A. Tyrosine kinase signaling pathways in neutrophils. Immunol Rev. 2016 Sep;273(1):121-39. doi: 10.1111/imr.12455. PMID 27558332
- [Background] Gilroy DW, Lawrence T, Perretti M, Rossi AG. Inflammatory resolution: new opportunities for drug discovery. Nat Rev Drug Discov. 2004 May;3(5):401-16. doi: 10.1038/nrd1383. No abstract available. PMID 15136788
- [Background] Hayes E, Pohl K, McElvaney NG, Reeves EP. The cystic fibrosis neutrophil: a specialized yet potentially defective cell. Arch Immunol Ther Exp (Warsz). 2011 Apr;59(2):97-112. doi: 10.1007/s00005-011-0113-6. Epub 2011 Feb 11. PMID 21311988
- [Background] Khan TZ, Wagener JS, Bost T, Martinez J, Accurso FJ, Riches DW. Early pulmonary inflammation in infants with cystic fibrosis. Am J Respir Crit Care Med. 1995 Apr;151(4):1075-82. doi: 10.1164/ajrccm/151.4.1075. PMID 7697234
- [Background] Koenderman L, Chilvers ER. Future treatment in patients with chronic obstructive pulmonary disease: to reverse or not to reverse steroid resistance-that is the question. J Allergy Clin Immunol. 2014 Aug;134(2):323-4. doi: 10.1016/j.jaci.2014.04.030. Epub 2014 Jun 13. No abstract available. PMID 24934274
- [Background] Laval J, Touhami J, Herzenberg LA, Conrad C, Taylor N, Battini JL, Sitbon M, Tirouvanziam R. Metabolic adaptation of neutrophils in cystic fibrosis airways involves distinct shifts in nutrient transporter expression. J Immunol. 2013 Jun 15;190(12):6043-50. doi: 10.4049/jimmunol.1201755. Epub 2013 May 20. PMID 23690474
- [Background] Leliefeld PH, Koenderman L, Pillay J. How Neutrophils Shape Adaptive Immune Responses. Front Immunol. 2015 Sep 14;6:471. doi: 10.3389/fimmu.2015.00471. eCollection 2015. PMID 26441976
- [Background] Mantovani A, Cassatella MA, Costantini C, Jaillon S. Neutrophils in the activation and regulation of innate and adaptive immunity. Nat Rev Immunol. 2011 Jul 25;11(8):519-31. doi: 10.1038/nri3024. PMID 21785456
- [Background] Martin C, Ohayon D, Alkan M, Mocek J, Pederzoli-Ribeil M, Candalh C, Thevenot G, Millet A, Tamassia N, Cassatella MA, Thieblemont N, Burgel PR, Witko-Sarsat V. Neutrophil-Expressed p21/waf1 Favors Inflammation Resolution in Pseudomonas aeruginosa Infection. Am J Respir Cell Mol Biol. 2016 May;54(5):740-50. doi: 10.1165/rcmb.2015-0047OC. PMID 26517580
- [Background] McKeon DJ, Condliffe AM, Cowburn AS, Cadwallader KC, Farahi N, Bilton D, Chilvers ER. Prolonged survival of neutrophils from patients with Delta F508 CFTR mutations. Thorax. 2008 Jul;63(7):660-1. doi: 10.1136/thx.2008.096834. No abstract available. PMID 18587042
- [Background] Meijer L, Nelson DJ, Riazanski V, Gabdoulkhakova AG, Hery-Arnaud G, Le Berre R, Loaec N, Oumata N, Galons H, Nowak E, Gueganton L, Dorothee G, Prochazkova M, Hall B, Kulkarni AB, Gray RD, Rossi AG, Witko-Sarsat V, Norez C, Becq F, Ravel D, Mottier D, Rault G. Modulating Innate and Adaptive Immunity by (R)-Roscovitine: Potential Therapeutic Opportunity in Cystic Fibrosis. J Innate Immun. 2016;8(4):330-49. doi: 10.1159/000444256. Epub 2016 Mar 18. PMID 26987072
- [Background] Moriceau S, Kantari C, Mocek J, Davezac N, Gabillet J, Guerrera IC, Brouillard F, Tondelier D, Sermet-Gaudelus I, Danel C, Lenoir G, Daniel S, Edelman A, Witko-Sarsat V. Coronin-1 is associated with neutrophil survival and is cleaved during apoptosis: potential implication in neutrophils from cystic fibrosis patients. J Immunol. 2009 Jun 1;182(11):7254-63. doi: 10.4049/jimmunol.0803312. PMID 19454722
- [Background] Moriceau S, Lenoir G, Witko-Sarsat V. In cystic fibrosis homozygotes and heterozygotes, neutrophil apoptosis is delayed and modulated by diamide or roscovitine: evidence for an innate neutrophil disturbance. J Innate Immun. 2010;2(3):260-6. doi: 10.1159/000295791. Epub 2010 Mar 10. PMID 20375556
- [Background] Ohayon D, De Chiara A, Chapuis N, Candalh C, Mocek J, Ribeil JA, Haddaoui L, Ifrah N, Hermine O, Bouillaud F, Frachet P, Bouscary D, Witko-Sarsat V. Cytoplasmic proliferating cell nuclear antigen connects glycolysis and cell survival in acute myeloid leukemia. Sci Rep. 2016 Oct 19;6:35561. doi: 10.1038/srep35561. PMID 27759041
- [Background] Peranzoni E, Zilio S, Marigo I, Dolcetti L, Zanovello P, Mandruzzato S, Bronte V. Myeloid-derived suppressor cell heterogeneity and subset definition. Curr Opin Immunol. 2010 Apr;22(2):238-44. doi: 10.1016/j.coi.2010.01.021. Epub 2010 Feb 17. PMID 20171075
- [Background] Pillay J, Kamp VM, van Hoffen E, Visser T, Tak T, Lammers JW, Ulfman LH, Leenen LP, Pickkers P, Koenderman L. A subset of neutrophils in human systemic inflammation inhibits T cell responses through Mac-1. J Clin Invest. 2012 Jan;122(1):327-36. doi: 10.1172/JCI57990. Epub 2011 Dec 12. PMID 22156198
- [Background] Pillay J, Ramakers BP, Kamp VM, Loi AL, Lam SW, Hietbrink F, Leenen LP, Tool AT, Pickkers P, Koenderman L. Functional heterogeneity and differential priming of circulating neutrophils in human experimental endotoxemia. J Leukoc Biol. 2010 Jul;88(1):211-20. doi: 10.1189/jlb.1209793. Epub 2010 Apr 16. PMID 20400675
- [Background] Pillay J, Tak T, Kamp VM, Koenderman L. Immune suppression by neutrophils and granulocytic myeloid-derived suppressor cells: similarities and differences. Cell Mol Life Sci. 2013 Oct;70(20):3813-27. doi: 10.1007/s00018-013-1286-4. Epub 2013 Feb 20. PMID 23423530
- [Background] Rossi AG, Sawatzky DA, Walker A, Ward C, Sheldrake TA, Riley NA, Caldicott A, Martinez-Losa M, Walker TR, Duffin R, Gray M, Crescenzi E, Martin MC, Brady HJ, Savill JS, Dransfield I, Haslett C. Cyclin-dependent kinase inhibitors enhance the resolution of inflammation by promoting inflammatory cell apoptosis. Nat Med. 2006 Sep;12(9):1056-64. doi: 10.1038/nm1468. Epub 2006 Sep 3. PMID 16951685
- [Background] Scapini P, Marini O, Tecchio C, Cassatella MA. Human neutrophils in the saga of cellular heterogeneity: insights and open questions. Immunol Rev. 2016 Sep;273(1):48-60. doi: 10.1111/imr.12448. PMID 27558327
- [Background] Uhel F, Azzaoui I, Gregoire M, Pangault C, Dulong J, Tadie JM, Gacouin A, Camus C, Cynober L, Fest T, Le Tulzo Y, Roussel M, Tarte K. Early Expansion of Circulating Granulocytic Myeloid-derived Suppressor Cells Predicts Development of Nosocomial Infections in Patients with Sepsis. Am J Respir Crit Care Med. 2017 Aug 1;196(3):315-327. doi: 10.1164/rccm.201606-1143OC. PMID 28146645
- [Background] Warbrick E. A functional analysis of PCNA-binding peptides derived from protein sequence, interaction screening and rational design. Oncogene. 2006 May 11;25(20):2850-9. doi: 10.1038/sj.onc.1209320. PMID 16407840
- [Background] Witko-Sarsat V. Neutrophils in the innate immunity conundrum of cystic fibrosis: a CFTR-related matter? J Innate Immun. 2013;5(3):195-6. doi: 10.1159/000350215. Epub 2013 Mar 23. No abstract available. PMID 23548924
- [Background] Witko-Sarsat V, Allen RC, Paulais M, Nguyen AT, Bessou G, Lenoir G, Descamps-Latscha B. Disturbed myeloperoxidase-dependent activity of neutrophils in cystic fibrosis homozygotes and heterozygotes, and its correction by amiloride. J Immunol. 1996 Sep 15;157(6):2728-35. PMID 8805680
- [Background] Witko-Sarsat V, Cramer EM, Hieblot C, Guichard J, Nusbaum P, Lopez S, Lesavre P, Halbwachs-Mecarelli L. Presence of proteinase 3 in secretory vesicles: evidence of a novel, highly mobilizable intracellular pool distinct from azurophil granules. Blood. 1999 Oct 1;94(7):2487-96. PMID 10498622
- [Background] Witko-Sarsat V, Halbwachs-Mecarelli L, Sermet-Gaudelus I, Bessou G, Lenoir G, Allen RC, Descamps-Latscha B. Priming of blood neutrophils in children with cystic fibrosis: correlation between functional and phenotypic expression of opsonin receptors before and after platelet-activating factor priming. J Infect Dis. 1999 Jan;179(1):151-62. doi: 10.1086/314532. PMID 9841834
- [Background] Witko-Sarsat V, Mocek J, Bouayad D, Tamassia N, Ribeil JA, Candalh C, Davezac N, Reuter N, Mouthon L, Hermine O, Pederzoli-Ribeil M, Cassatella MA. Proliferating cell nuclear antigen acts as a cytoplasmic platform controlling human neutrophil survival. J Exp Med. 2010 Nov 22;207(12):2631-45. doi: 10.1084/jem.20092241. Epub 2010 Oct 25. PMID 20975039
- [Background] Witko-Sarsat V, Ohayon D. Proliferating cell nuclear antigen in neutrophil fate. Immunol Rev. 2016 Sep;273(1):344-56. doi: 10.1111/imr.12449. PMID 27558345
- [Background] Witko-Sarsat V, Pederzoli-Ribeil M, Hirsch E, Sozzani S, Cassatella MA. Regulating neutrophil apoptosis: new players enter the game. Trends Immunol. 2011 Mar;32(3):117-24. doi: 10.1016/j.it.2011.01.001. Epub 2011 Feb 12. PMID 21317039
- [Background] Witko-Sarsat V, Rieu P, Descamps-Latscha B, Lesavre P, Halbwachs-Mecarelli L. Neutrophils: molecules, functions and pathophysiological aspects. Lab Invest. 2000 May;80(5):617-53. doi: 10.1038/labinvest.3780067. No abstract available. PMID 10830774
- [Background] Witko-Sarsat V, Sermet-Gaudelus I, Lenoir G, Descamps-Latscha B. Inflammation and CFTR: might neutrophils be the key in cystic fibrosis? Mediators Inflamm. 1999;8(1):7-11. doi: 10.1080/09629359990658. PMID 10704083
- [Background] Worlitzsch D, Tarran R, Ulrich M, Schwab U, Cekici A, Meyer KC, Birrer P, Bellon G, Berger J, Weiss T, Botzenhart K, Yankaskas JR, Randell S, Boucher RC, Doring G. Effects of reduced mucus oxygen concentration in airway Pseudomonas infections of cystic fibrosis patients. J Clin Invest. 2002 Feb;109(3):317-25. doi: 10.1172/JCI13870. PMID 11827991
- [Background] Wright HL, Makki FA, Moots RJ, Edwards SW. Low-density granulocytes: functionally distinct, immature neutrophils in rheumatoid arthritis with altered properties and defective TNF signalling. J Leukoc Biol. 2017 Feb;101(2):599-611. doi: 10.1189/jlb.5A0116-022R. Epub 2016 Sep 6. PMID 27601627
- [Background] Heijerman HGM, McKone EF, Downey DG, Van Braeckel E, Rowe SM, Tullis E, Mall MA, Welter JJ, Ramsey BW, McKee CM, Marigowda G, Moskowitz SM, Waltz D, Sosnay PR, Simard C, Ahluwalia N, Xuan F, Zhang Y, Taylor-Cousar JL, McCoy KS; VX17-445-103 Trial Group. Efficacy and safety of the elexacaftor plus tezacaftor plus ivacaftor combination regimen in people with cystic fibrosis homozygous for the F508del mutation: a double-blind, randomised, phase 3 trial. Lancet. 2019 Nov 23;394(10212):1940-1948. doi: 10.1016/S0140-6736(19)32597-8. Epub 2019 Oct 31. PMID 31679946